CLINICAL TRIAL: NCT04182490
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Single Dose Regimen Study of LMN-101 in Healthy Volunteers Challenged With Campylobacter Jejuni
Brief Title: LMN-101 in a Campylobacter Human Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumen Bioscience, Inc. (Industry)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Pharmaron (Industry); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAM02
Record Dates: First submitted 2019-09-19; First posted 2019-12-02 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Campylobacter Infections
MeSH Terms: conditions — Campylobacter Infections | interventions — Starch

STUDY DESIGN:
Intervention Model Description: Healthy adults are treated with LMN-101 or placebo followed by an oral challenge of campylobacter to compare the frequency of solicited and unsolicited adverse events in subjects that received LMN-101 compared to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical-appearing placebo capsules, pharmacy blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3000-mg cohort (Active Comparator): LMN-101, six 500-mg capsules orally three times daily for 14 days (n=21)
  Interventions: Biological: LMN-101
- Placebo cohort (Placebo Comparator): Placebo, six 500-mg capsules orally three times daily for 14 days (n=21)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: LMN-101 — VHH-derived binding protein designed to bind and inhibit FlaA, flagellin filament protein of Campylobacter jejuni, delivered in whole spray-dried, spirulina biomass
  Other Names: Variable heavy chain (VHH) binding protein against flagellin
  Arms: 3000-mg cohort
Drug: Placebo — Identical appearing placebo
  Other Names: Corn starch
  Arms: Placebo cohort

SUMMARY:
Randomized, double-blind, placebo-controlled, single dose regimen study of LMN-101 followed by Campylobacter jejuni challenge. Subjects will initially, after documentation of informed consent, begin taking their assigned LMN-101 or placebo regimen three times daily. After two days, subjects will receive the C. jejuni challenge inoculum. Subjects will begin an appropriate antibiotic course upon meeting early treatment criteria or 144 hours following C. jejuni challenge, whichever is earlier. Subjects will be allowed to leave the clinical research facility 3 days after antibiotics, when all symptoms have resolved or are resolving, and have had ≥ 2 consecutive stool cultures ≥ 12 hours apart negative for C. jejuni and are afebrile > 24 hours prior to release and off antipyretics within 24 hours of discharge. Subjects will continue taking their LMN-101 or placebo regimen three times daily for a total of 14 days. Subjects will be provided a diary card/memory aid and thermometer for at-home monitoring of solicited adverse events through Day 24. Subjects will be seen at research facility for protocol-specified evaluations and will also be contacted by telephone 6 months after challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female between 18 and 50 years of age, inclusive, at time of informed consent
2. Willingness to participate after written informed consent obtained
3. Available for all planned clinical visits (for physical examinations, blood draws, and stool collections) and follow-up monitoring (9 or 10 clinic visits and 1 phone interview 6 months post-challenge)
4. Agreement to follow the restrictions of the study. Willing and able to follow the study directions and procedures, including the rules and procedures of the clinical research unit.
5. Demonstrated comprehension of the protocol procedures including knowledge of Campylobacter illness by passing a written examination (passing grade ≥ 70%).
6. General good health, without significant medical illness or abnormal physical examination findings as determined by the PI.
7. Laboratory values are Grade 1 or lower using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 as defined below:

   1. Absolute neutrophil count ≥ 1500/μL
   2. Lymphocyte count ≥ 800/μL
   3. Platelet count ≥ 125,000/μL
   4. Hemoglobin ≥ 13.0 g/dL in males (≥ 11.0 g/dL in females)
   5. Serum creatinine ≤1.5x ULN
   6. ALT and/or AST ≤ 1.5x ULN
   7. Total bilirubin ≤ 1.5x ULN
8. Females of childbearing potential must commit to use one of the following highly effective methods of birth control consistently for at least 1 month prior to screening through study completion:

   1. Stable hormonal contraception with inhibition of ovulation; or
   2. Intrauterine device (IUD); or
   3. Bilateral tubal occlusion; or
   4. Surgical sterilization (vasectomy) of male partner at least 6 months prior to study; or
   5. Sexual abstinence (inactivity).
9. To be considered of non-childbearing potential, females should be surgically sterilized (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be post-menopausal and at least 1 year since menses with follicle-stimulating hormone ≥ 40 units.
10. Males should use condoms for contraception and refrain from donating sperm through Day 64.
11. BMI between 18.5 and 33.5 inclusive
12. Complies with current Pharmaron Covid-19 policies and procedures

Exclusion Criteria

1. Significant medical condition or laboratory abnormalities that in the opinion of the Principal Investigator preclude participation in the study.
2. History of Covid symptoms or positive Covid test within 2 weeks prior to admission date.
3. Alcohol or illicit drug abuse/dependency
4. Positive serology results for HIV, HBsAg, or HCV with confirmatory assays.
5. Pregnancy or breastfeeding
6. Personal or documented family history of Guillain-Barr syndrome or neuromuscular disease; or an inflammatory arthritis such as reactive arthritis, ankylosing spondylitis, or rheumatoid arthritis; inflammatory bowel disease; autoimmune disease; malignancy (not including basal cell carcinoma); any immunocompromising condition; or history of major gastrointestinal surgery.
7. Evidence of neurological abnormalities.
8. History of reactive arthritis or evidence of inflammatory arthritis on exam.
9. Fever within the 2 weeks prior to time of enrollment.
10. Evidence of IgA deficiency (serum IgA < 7 mg/mL or below the limit of detection of assay).
11. HLA-B27 positive
12. Allergy or prior intolerance to two or more of the following antibiotics: azithromycin, ciprofloxacin, levofloxacin, erythromycin, ampicillin, or amoxicillin/clavulanate.
13. Allergy or prior intolerance to spirulina or spirulina products.
14. Fewer than 3 stools per week or more than 3 stools per day as the usual frequency.
15. History of moderate to serious diarrhea while traveling in a developing country within the last 3 years.
16. History of myocarditis or pericarditis.
17. History of major abdominal surgery or unexplained abdominal scar. Ok if appendectomy or cholecystectomy (one year post)
18. Regular use of antidiarrheal, antacids, loperamide, bismuth subsalicylate diphenoxylate, or similar medication affecting bowel motility (regular defined as at least weekly).
19. Use of proton pump inhibitors, H2 blockers, or other antacids within 48 hours preceding initiation of LMN-101 or placebo.
20. Use of antibiotics during the 7 days preceding initiation of LMN-101 or placebo.
21. Use of spirulina, or spirulina containing products, other than the study drug in the 30 days preceding initiation of LMN-101 or placebo.
22. Use of any investigational product within 30 days preceding initiation of LMN-101 or placebo or planned use during the active study period.
23. Use of any medication known to affect the immune system (e.g., systemic corticosteroids, chemotherapy, monoclonal antibody biologic response modifiers) within 12 months preceding initiation of LMN-101 or placebo or planned use during the active study period (excluding inhaled steroids with spacer).
24. History of prior exposure to Campylobacter including by vaccination or infection in previous trials, or serum immunoglobulin A (IgA) titer to C. jejuni glycine extract >1:4000.
25. Other dietary or environmental exposures that may place the subject at high risk for prior Campylobacter exposure (to be determined on a case-by-case basis by the PI).
26. Employment as a food handler; childcare worker; or caregiver for elderly, immunocompromised individuals, or other at-risk population.
27. History of major mental illness such as schizophrenia, major depression or suicidal ideation
28. Any other criteria which, in the Principal Investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study or the results of the study.
29. Potential participant's 12 - lead electrocardiogram demonstrating pathologic abnormalities including non-sinus rhythm, pathologic Q waves, significant ST-T wave changes, corrected QT interval (QTc) using Fridericia correction (QTcF) at screening and Day -1 (admission) >450 msec.
30. At screening, systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MB,ChB, FACP, Principal Investigator — Pharmaron
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3000-mg Cohort | Placebo Cohort
Started | 21 | 21
Completed | 18 | 16
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: 42 healthy volunteers
Groups:
- Total: Total of all reporting groups
Arm/Group | 3000-mg Cohort | Placebo Cohort | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (7.74) | 32.8 (9.51) | 33.4 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 12 | 28
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited or Unsolicited Adverse Events
Description: Number of participants with solicited or unsolicited adverse events that received LMN-101 compared to placebo for the protocol-specified duration of collection for each type of adverse event.
Time Frame: Day 1 to Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | 3000-mg Cohort | Placebo Cohort
Number analyzed (Participants) | 21 | 21
Participants
  Solicited Adverse Events | 15 | 16
  Unsolicited Adverse Events | 17 | 16

ADVERSE EVENTS:
Time Frame: 59 Days
Arm/Group | 3000-mg Cohort | Placebo Cohort
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 20/21 | 18/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3000-mg Cohort (N=21) | Placebo Cohort (N=21)
Diarrhea (Gastrointestinal disorders) | 19 (21) | 14 (16)
Abdominal Pain (Gastrointestinal disorders) | 15 (29) | 14 (23)
Nausea (Gastrointestinal disorders) | 8 (8) | 7 (7)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 15 (21) | 12 (19)
Chills (General disorders) | 12 (13) | 12 (13)
Pyrexia (General disorders) | 12 (14) | 8 (8)
Fatigue (General disorders) | 11 (12) | 9 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Tachycardia (Cardiac disorders) | 8 (8) | 5 (5)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Neutrophil count increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Differential white blood cell count abnormal (Investigations) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dizzyness (Nervous system disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT04182490/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT04182490/SAP_001.pdf